CLINICAL TRIAL: NCT01965275
Title: An Open,Multi Center Trial to Evaluate the Efficacy and Safety of High-Dose,Pulsatile Erlotinib/Gefitinib for Advanced Non-Small Cell Lung Cancer Patients After Failure of Standard Dose EGFR-TKIs
Brief Title: High-Dose,Pulsatile Erlotinib/Gefitinib for Advanced NSCLC Patients After Failure of Standard Dose EGFR-TKIs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Pan Yueyin, Professor, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDP-ADNSCLC
Record Dates: First submitted 2013-10-10; First posted 2013-10-18 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Self Efficacy; Drug Toxicity
Keywords: Advanced non-small cell lung cancer; High-dose; Pulsatile; EGFR-TKIs
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib or Gefitinib (Experimental): Patients received the treatment with high-dose, pulsatile Erlotinib(600 mg every 4 days) or Gefitinib (1000 mg every 4 days) until disease progression or unacceptable toxicity occurred. The overall study period takes about 12 months
  Interventions: Drug: Erlotinib or Gefitinib

INTERVENTIONS:
Drug: Erlotinib or Gefitinib — Patients received the treatment with high-dose, pulsatile Erlotinib(600 mg every 4 days) or Gefitinib (1000 mg every 4 days) until disease progression or unacceptable toxicity occurred. The overall study period takes about 12 months
  Other Names: high-dose, pulsatile Erlotinib or Gefitinib

SUMMARY:
the purpose of this study is to evaluate the efficacy and safety of high-dose，pulsatile Erlotinib/Gefitinib in advanced non small cell lung cancer (NSCLC) patients after failure of standard dose EGFR-TKIs（Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitors）

DETAILED DESCRIPTION:
To evaluate the efficacy and safety by treating the advanced non small cell lung cancer (NSCLC) patients who have failure of standard dose EGFR-TKIs(Erlotinib or Gefitinib ) with high-dose, pulsatile Erlotinib(450mg every 3 days) or Gefitinib (1000mg every 4 days)

ELIGIBILITY:
Inclusion Criteria:

* 1. NSCLC patients were confirmed by histology or cytology 2. Patients were ever treated with standard dose EGFR-TKIs(Erlotinib or Gefitinib )on which he/she achieved complete remission/partial remission,or maintained stable disease for 4 months.Disease progression at present (accord to RECISTv1.1 criteria） 3.At least one target lesion that has not previously been radiated and is measurable according to RECIST v1.1; 4.Have an ECOG PS of 0-2 5.At least 8 weeks of expected survival time 6.Have no serious cardiovascular,hepatobiliary or renal disorders 7.Provision of a voluntarily given, personally signed and dated, written informed consent document 8.Must be in accordance with the following laboratory biochemical data: Hgb≥80g/L，WBC≥3.0×10^9/L，ANC≥1.0×10^9/L， PLT≥80×10^9/L Renal function：SCr≤ULN Liver function： if no hepatic metastases:AST/ALT≤2.5ULN if hepatic metastases:AST/ALT≤5ULN

Exclusion Criteria:

* If the subject meet any of the following exclusion criteria ,he/she is no eligible to participate in this study

  1. Have chronic toxicity reaction(above grade 2) and not recovered( hair loss not include)
  2. Have Appeared skin rashes or diarrhea(above grade 3),or have any reason lead to decrement during standard dose EGFR-TKIs treatment
  3. Female subjects who are in pregnancy or lactation，or of childbearing age but don't take any contraceptive measures
  4. Current enrollment in another therapeutic clinical study
  5. Have any symptoms of brain metastases or leptomeningeal metastases
  6. Subjects will not be eligible if they have history of prior malignancy in past 5 years
  7. Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this study or known drug abuse/alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
efficacy and safety | 1 year
  To evaluate the efficacy and safety by treating the advanced NSCLC patients who have failure of standard dose EGFR-TKIs with high-dose, pulsatile Erlotinib(600mg every 4 days) or Gefitinib (1000mg every 4 days)
  Radiologically measurable disease by RECIST v1.1 criteria:
  1. At least one target lesion that has not previously been radiated and is measurable according to RECIST v1.1;
  2. Acceptable radiologic procedures for disease assessment include contrast enhanced conventional or spiral computed tomography (CT), or contrast enhanced magnetic resonance imaging (MRI); Non-contrast CT scan is acceptable only for subjects who are both allergic to intravenous contrast and unable to cooperate with MRI, or MRI is not available. The following are not allowed as sole documentation of target lesions: CT component of a positron emission tomography (PET)/CT,ultrasound alone, nuclear scans (including bone or PET scans), chest X-ray or bone radiographs, and tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: Yueyin Pan, PHD,MD, Principal Investigator — Anhui Medical University
Locations (1):
- Dept. of Oncology,The First Affiliated Hospital of Anhui Medical Univesrsity, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided